CLINICAL TRIAL: NCT00640341
Title: Product Performance of Bausch & Lomb PureVision® Contact Lens When Compared to Johnson & Johnson Acuvue Oasys Contact Lens and the Ciba Vision O2Optix Contact Lens Worn Daily.
Brief Title: Comparative Performance of PureVision, Acuvue Oasys and O2Optix
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 552
Record Dates: First submitted 2008-02-20; First posted 2008-03-21 (Estimated); Results first posted 2011-03-31 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- PureVision (Experimental): PureVision Contact Lens
  Interventions: Device: PureVision Contact Lens
- Acuvue Oasys (Active Comparator): Acuvue Oasys Contact Lens
  Interventions: Device: Acuvue Oasys Contact Lens
- O2Optix (Active Comparator): O2Optix Contact Lens
  Interventions: Device: O2Optix Contact lens

INTERVENTIONS:
Device: PureVision Contact Lens — contact lens for daily wear
  Arms: PureVision
Device: Acuvue Oasys Contact Lens — contact lens for daily wear
  Arms: Acuvue Oasys
Device: O2Optix Contact lens — contact lens for daily wear
  Arms: O2Optix

SUMMARY:
The objective of this study is to evaluate the performance of the PureVision Contact Lens compared to Acuvue Oasys Contact lens and O2Optix Contact lens when worn on a daily wear basis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is myopic
* VA correctable to 0.3 LogMAR or better (driving vision)
* Clear central cornea
* Subject uses a lens care system on a regular basis

Exclusion Criteria:

* Systemic disease affecting ocular health
* Using systemic or topical medications
* Wear monovision, multifocal or toric contact lenses
* Any grade 2 or greater slit lamp findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Cairns, MCOptom, PhD, Study Director — Bausch & Lomb Incorporated; Bruce Anderson, OD, Principal Investigator — Anderson & Associates
Locations (1):
- Anderson & Associates, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 546 subjects (1092 eyes) were planned to be enrolled at 26 investigative sites in the US. First subject enrolled on 2/25/2008 and last subject seen was 4/28/2008.
Pre-assignment Details: 510 subjects (1020 eyes) were enrolled (all were dispensed). 477 subjects (954 eyes) completed the study. 10 subjects were ineligible at baseline and 23 were discontinued during the study.
Groups:
- PureVision: Redesigned PureVision Contact Lens. Lenses are to be worn on a daily wear basis.
- Acuvue Oasys: Currently marketed Acuvue Oasys Contact Lens. Lenses are to be worn on a daily wear basis.
- O2Optix: Currently marketed O2Optix Contact Lens. Lenses are to be worn on a daily wear basis.
Period: Overall Study
Arm/Group | PureVision | Acuvue Oasys | O2Optix
Started | 170 (All Starting participants were dispensed lenses) | 170 | 170
Eligible Participants at Baseline | 165 | 167 | 168
Completed | 149 | 165 | 163
Not Completed | 21 | 5 | 7
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Positive Slit Lamp Findings | 0 | 0 | 1
Not completed — Study Related Symptoms/Complaints | 2 | 1 | 2
Not completed — Inability to Maintain Wearing Schedule | 1 | 1 | 0
Not completed — Failure to Follow Subject Instructions | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 1
Not completed — Unacceptable Lens Movement | 1 | 0 | 0
Not completed — Poor fit/Uncomfortable | 4 | 0 | 0
Not completed — Ineligable at Baseline | 5 | 3 | 2
Not completed — Adverse event and positive slit lamp | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PureVision | Acuvue Oasys | O2Optix | Total
Number analyzed (Participants) | 165 | 167 | 168 | 500
Age, Customized [Number; unit: Participants]
  Age 18 to 65 years | 165 | 167 | 168 | 500
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 127 | 124 | 376
  Male | 40 | 40 | 44 | 124
Region of Enrollment [Number; unit: Participants]
  United States | 165 | 167 | 168 | 500

OUTCOME MEASURES:

1. Primary Outcome: Any Slit Lamp Finding > Grade 2
Description: All dispensed eyes over all follow-up visits. Measured on a scale of 0-4 with 0=no findings and 4=severe findings. Epithelial edema, epithelial microcysts, corneal staining, limbal & bulbar injection, conjunctival abnormalities, corneal neovascularization and infiltrates were measured.
Time Frame: Over all follow-up visits for the 1 month study period
Population: All dispensed eyes
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | PureVision | Acuvue Oasys | O2Optix
Number analyzed (Participants) | 162 | 169 | 168
Number analyzed (eyes) | 324 | 338 | 336
Eyes | 2 | 5 | 10

2. Primary Outcome: Subjective Responses to Comfort-related Symptoms/Complaints
Description: Subjective ratings of symptoms/complaints using a scale of 0 = Severe Stinging/Burning to 100 = No Stinging/Burning for each eye; 0 represented the least favorable rating and a 100 represented the most favorable rating.
Time Frame: Over all follow-up visits for 1 month study period
Population: All eligible dispensed eyes.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: eyes
Arm/Group | PureVision | Acuvue Oasys | O2Optix
Number analyzed (Participants) | 157 | 167 | 164
Number analyzed (eyes) | 314 | 334 | 328
Units on a Scale
  Morning Comfort | 85.5 (17.55) | 92.9 (11.97) | 92.0 (12.79)
  Comfort Throughout the Day | 82.9 (18.94) | 90.1 (14.47) | 88.4 (13.43)
  End of Day Comfort | 76.1 (21.86) | 85.2 (16.69) | 81.4 (18.40)
  Lens Awareness | 79.9 (23.46) | 89.5 (16.30) | 86.4 (17.91)
  Irritation | 81.7 (20.15) | 90.5 (14.42) | 87.0 (15.89)
  Itching | 89.9 (15.75) | 93.5 (12.81) | 92.2 (13.57)
  Dryness | 81.9 (20.22) | 89.1 (14.42) | 85.0 (17.46)
  Redness | 91.0 (14.93) | 94.5 (11.14) | 91.9 (14.23)

3. Primary Outcome: Uncorrected Distance High Contrast Visual Acuity
Description: logMAR high contrast visual acuity (VA) over all visits.
Time Frame: Over all visits for the 1 month study period
Population: All eligible dispensed eyes.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | PureVision | Acuvue Oasys | O2Optix
Number analyzed (Participants) | 164 | 167 | 168
Number analyzed (eyes) | 328 | 334 | 336
LogMAR | -0.031 (0.070) | -0.026 (0.071) | -0.024 (0.0760)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | PureVision | Acuvue Oasys | O2Optix
Serious Adverse Events (participants affected / at risk) | 0/340 | 0/340 | 0/340
Other Adverse Events (participants affected / at risk) | 0/340 | 0/340 | 0/340

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.